CLINICAL TRIAL: NCT00713323
Title: A Multicentre, Open Label, Follow on Study to Assess the Maintenance of Effect, Tolerance and Safety of Sativex® in the Treatment of Subjects With Neuropathic Pain. This Will be Followed by a Randomised-withdrawal Phase (Part B) for a Subset of Patients.
Brief Title: A Study to Compare the Safety and Tolerability of Sativex® in Patients With Neuropathic Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GWCL0404 Part A
Record Dates: First submitted 2008-07-10; First posted 2008-07-11 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Pain; Peripheral Neuropathy
Keywords: Pain; Peripheral Neuropathy
MeSH Terms: conditions — Pain; Peripheral Nervous System Diseases | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sativex (Experimental): Active treatment
  Interventions: Drug: Sativex®

INTERVENTIONS:
Drug: Sativex® — containing THC (27 mg/ml):CBD (25 mg/ml), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Maximum permitted dose was eight actuations in any three hour period and 24 actuations (THC 65 mg: CBD 60 mg) in 24 hours
  Other Names: GW-1000-02

SUMMARY:
The purpose of this study is to assess the safety and tolerability of long term therapy with Sativex® in relieving neuropathic pain.

DETAILED DESCRIPTION:
This was a 38 week, multicentre, open label (Part A) follow-on study to evaluate, the maintenance of effect of, the development of tolerance through exposure to, and safety of, Sativex® in the treatment of subjects with neuropathic pain. The study provided continued availability of Sativex® to subjects who completed the preceding double-blind neuropathic pain studies. Consenting, eligible subjects who had participated in previous GW Pharma Ltd (GW) randomised, placebo-controlled clinical studies entered the study (Visit 1, Day 0) and commenced dosing. Study visits took place at Week 2 (Visit 2, Day 14), Week 14 (Visit 3, Day 98), and Week 26 (Visit 4, Day 182). Subjects returned to the centre for an end of treatment visit at week 38 (Visit 5, Day 266). All subjects received Sativex®. This was followed by a five week randomised-withdrawal phase (Part B) for a subset of subjects. An end of study visit took place 28 days after Visit 5 (or 5b or 5c) or withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* Had participated in a GW clinical study to investigate the effects of Sativex® on peripheral neuropathic pain and had completed the study. This must have been within the last seven days
* Had complied with all of the study requirements in the preceding GW parent RCTs, including the completion of diary cards and study questionnaires
* Had shown tolerability to the study medication in a preceding GW study
* Was expected, in the opinion of the investigator, to gain clinical benefit from receiving Sativex® therapy
* Ability (in the investigators opinion) and willingness to comply with all study requirements, including the completion of diary cards and study questionnaires
* Agreement for the responsible authorities (as applicable in individual countries), their primary care physician, and their consultant, if appropriate, to be notified of their participation in the study.

Exclusion Criteria:

* History of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition
* Known or suspected history of alcohol or substance abuse
* History of epilepsy or recurrent seizures
* Known or suspected hypersensitivity to cannabinoids or any of the excipients of the study medication Evidence of cardiomyopathy
* Experienced myocardial infarction or clinically relevant cardiac dysfunction within the last 12 months or had a cardiac disorder that, in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction
* QT interval; of > 450 ms (males) or > 470 ms (females) at Visit 1
* Secondary or tertiary AV block or sinus bradycardia (HR <50bpm unless physiological) or sinus tachycardia (HR>110bpm) at Visit 1
* Diastolic blood pressure of <50 mmHg or >105 mmHg in a sitting position at rest for five minutes prior to measurement at Visit 1
* Impaired renal function i.e., creatinine clearance is lower than 50ml/min at Visit 1 and is indicative of renal impairment
* Significantly impaired hepatic function, at Visit 1, in the Investigator's opinion
* Female subjects of child bearing potential and male subjects whose partner was of child bearing potential, unless they were willing to ensure that they or their partner used effective contraception during the study and for three months thereafter
* If female, were pregnant or lactating, or were planning pregnancy during the course of the study and for three months thereafter
* Received an IMP within the 12 weeks before Visit 1 (except the prerequisite study medication from the GW parent RCTs)
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, may influence the result of the study or the subject's ability to participate in the study
* Following a physical examination, the subject had any abnormalities that, in the opinion of the investigator, would prevent the subject from safely participating in the study.
* Intention to donate blood during the study
* Previous randomisation into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2005-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hoggart, MBBS, FRCA, Principal Investigator — Pain Management Research, Clinical Trials Unit, Netherwood House, Solihull Hospital
Locations (1):
- Pain Management Research, Clinical Trials Unit, Netherwood House, Solihull Hospital, Solihull, West Midlands, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex: Subjects received Sativex delivered in 100 μl actuations by a pump action oromucosal spray. Maximum permitted dose was 24 actuations in 24 hours (THC 65 mg:CBD 60 mg).
Period: Overall Study
Arm/Group | Sativex
Started | 380
Completed | 234
Not Completed | 146
Not completed — Adverse Event | 75
Not completed — Withdrawal by Subject | 15
Not completed — Lost to Follow-up | 11
Not completed — Lack of Efficacy | 36
Not completed — Low creatine clearance at screening | 1
Not completed — Withdrawn due to exclusion criteria 11 | 1
Not completed — Surgery cured allodynic pain | 1
Not completed — Pain free | 1
Not completed — Non-compliance | 1
Not completed — Pain resolved | 1
Not completed — Subject travelling to USA | 1
Not completed — Subject travelling to Dominica Republic | 1
Not completed — Treatment that may interact with Sativex | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sativex
Number analyzed (Participants) | 380
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 287
  >=65 years | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180
  Male | 200
Region of Enrollment [Number; unit: participants]
  United Kingdom | 222
  Belgium | 9
  Canada | 5
  Romania | 50
  Czech Republic | 94

OUTCOME MEASURES:

1. Primary Outcome: Change From Parent Study Baseline in Mean Pain 0-10 Numerical Rating Scale (NRS) Score During the Last 4 Weeks of Open-label Treatment
Description: The average pain NRS was complete at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your pain or average pain in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of pain. A negative value indicates an improvement in pain score from baseline.
Time Frame: 38 weeks
Population: All subjects who received at least one dose of open-label Sativex were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex
Number analyzed (Participants) | 365
units on a scale | -2.07 (2.13)

2. Secondary Outcome: Change From Parent Study Baseline in Mean Neuropathic Pain Scale (NPS) Score at End of Open-label Treatment (Week 38)
Description: The NPS score is 0-100 sum of 10 individual pain scores (0-10 NRS, 0= no pain to 10 = most pain imaginable). A negative change from baseline indicates an improvement in pain.
Time Frame: 38 weeks
Population: All subjects who received at least one dose of open-label Sativex were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex
Number analyzed (Participants) | 371
units on a scale | -15.67 (19.11)

3. Secondary Outcome: Change From Parent Study Baseline in Mean Sleep Quality 0-10 NRS Score at the End of Open-label Treatment (Week 38)
Description: The sleep disruption NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate how your pain disrupted your sleep last night?" where 0 = did not disrupt sleep and 10 = completely disrupted (unable to sleep at all). A negative value indicates an improvement in sleep disruption score from baseline.
Time Frame: 38 weeks
Population: All subjects who received at least one dose of open-label Sativex were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex
Number analyzed (Participants) | 374
units on a scale | -1.76 (2.93)

4. Secondary Outcome: Subject Global Impression of Change
Description: A 7-point Likert-type scale was used, with the question: 'Please assess the status of your pain since entry into the study using the scale below' with the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse or very much worse". At Visit 2 (Baseline) patients wrote a brief description of their pain which was used at Week 5 to aid their memory regarding their symptoms at study start. For each of above markers the number of participants were reported.
Time Frame: week 38
Population: All subjects who received at least one dose of open-label Sativex were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Sativex
Number analyzed (Participants) | 380
participants
  Very Much Improved | 41
  Much Improved | 107
  Slightly Improved | 99
  No change | 79
  Slightly worse | 14
  Much worse | 12
  Very much worse | 4
  Missing Information | 24

5. Secondary Outcome: Change From Parent Study Baseline in Mean EuroQol-5D Weighted Health State Index Score at the End of Open-label Treatment
Description: The EQ-5D questionnaire provided two outcomes:(1)A weighted health state index visual analogue scale (VAS); (2) A self-rated health status VAS. EQ-5D Health Status VAS Scale: 0 = worst health state imaginable to 100 = best health state imaginable. An increase in score indicates an improvement in condition.The weighted health state index used the same VAS as above but was calculated for each assessment without imputation to account for missing values i.e., if one or more individual items was missing then the whole index was missing.
Time Frame: 38 weeks
Population: All subjects who received at least one dose of open-label Sativex were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex
Number analyzed (Participants) | 380
units on a scale | 0.07 (0.208)

6. Secondary Outcome: Change From Parent Study Baseline in Mean EuroQol-5D Self-rated Health Status Visual Analogue Scale Score at the End of Open-label Treatment
Description: The EQ-5D questionnaire provided two outcomes:(1)A weighted health state index visual analogue scale (VAS); (2) A self-rated health status VAS. EQ-5D Health Status VAS Scale: 0 = worst health state imaginable to 100 = best health state imaginable. An increase in score indicates an improvement in condition.
Time Frame: 38 weeks
Population: All subjects who received at least one dose of open-label Sativex were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex
Number analyzed (Participants) | 380
units on a scale | 6.27 (23.35)

7. Secondary Outcome: Incidence of Adverse Events as a Measure of Subject Safety
Description: The number of subjects who reported an adverse event during Part A of the study is presented (including the follow-up period of 28 days following cessation of opel-label treatment).
Time Frame: 42 weeks
Population: All subjects who received at least one dose of open-label Sativex were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Sativex
Number analyzed (Participants) | 380
participants | 295

8. Secondary Outcome: Change From Parent Study Baseline in Mean Intoxication 0-10 Numerical Rating Scale Score at the End of Open-label Treatment (38 Weeks)
Description: The patient was asked "on a scale of '0 to 10' please indicate the average level of your intoxication due to medications over the last 24 hours" (0=no intoxication and 10=extreme toxication). A negative value indicates an improvement in pain score from baseline.
Time Frame: 38 weeks
Population: All subjects who received at least one dose of open-label Sativex were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex
Number analyzed (Participants) | 356
units on a scale | 0.6 (2.62)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring from the time of consent to post study follow up i.e. 42 weeks were collected. All deaths and serious adverse events (SAEs) occurring within 28 days of the final dose of open-label treatment were also collected.
Description: All AEs occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex
Serious Adverse Events (participants affected / at risk) | 40/380
Other Adverse Events (participants affected / at risk) | 295/380
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=380)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 2
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1
INTESTINAL FUNCTIONAL DISORDER (Gastrointestinal disorders) | 1
OESOPHAGEAL DISCOMFORT (Gastrointestinal disorders) | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
CHEST PAIN (General disorders) | 2
OEDEMA PERIPHERAL (General disorders) | 2
PYREXIA (General disorders) | 1
CELLULITIS (Infections and infestations) | 2
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 2
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1
LOCALISED INFECTION (Infections and infestations) | 1
ORAL FUNGAL INFECTION (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
HEPATIC ENZYME INCREASED (Investigations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEURILEMMOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
AMNESIA (Nervous system disorders) | 2
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
CERVICAL ROOT PAIN (Nervous system disorders) | 1
DIABETIC COMA (Nervous system disorders) | 1
FACIAL PARESIS (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 1
PARAPLEGIA (Nervous system disorders) | 1
SOMNOLENCE (Nervous system disorders) | 1
SPINAL CORD INFARCTION (Nervous system disorders) | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
DISORIENTATION (Psychiatric disorders) | 1
PARANOIA (Psychiatric disorders) | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
PELVIC PAIN (Reproductive system and breast disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 2
HYPERTENSION (Vascular disorders) | 1
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 1
THROMBOPHLEBITIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=380)
Dizziness (Nervous system disorders) | 79
Dysgeusia (Nervous system disorders) | 29
Somnolence (Nervous system disorders) | 28
Headache (Nervous system disorders) | 23
Balance Disorder (Nervous system disorders) | 12
Memory Impairment (Nervous system disorders) | 12
Nausea (Gastrointestinal disorders) | 42
Dry Mouth (Gastrointestinal disorders) | 30
Vomiting (Gastrointestinal disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 17
Mouth Ulceration (Gastrointestinal disorders) | 16
Fatigue (General disorders) | 31
Feeling Drunk (General disorders) | 21
Nasopharyngitis (Infections and infestations) | 15
Urinary Tract Infection (Infections and infestations) | 13
Disorientation (Psychiatric disorders) | 19
Depressed Mood (Psychiatric disorders) | 13
Insomnia (Psychiatric disorders) | 13
Depression (Psychiatric disorders) | 12
Dissociation (Psychiatric disorders) | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 10
Hypoglycaemia (Metabolism and nutrition disorders) | 12
Accident (Injury, poisoning and procedural complications) | 11
Hypertension (Vascular disorders) | 10
Vertigo (Ear and labyrinth disorders) | 14
Lower Respiratory Tract Infection (Infections and infestations) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.